CLINICAL TRIAL: NCT01019733
Title: Intrathecal Autologous Stem Cells for Children With Hipoxic/Ischemic Brain Injury
Brief Title: Intrathecal Stem Cells in Brain Injury
Acronym: ISC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Maria del Consuelo Mancías Guerra, Hospital Universitario Dr. José E. González
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE09-014
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Hypoxia-Ischemia, Cerebral; Cerebral Palsy
Keywords: Hypoxia; Ischemia; Brain; Children; Cerebral Palsy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Cerebral Palsy; Hypoxia; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients (Experimental): Children whom will receive intrathecal autologous stem cells
  Interventions: Procedure: Intrathecal Autologous Stem Cells

INTERVENTIONS:
Procedure: Intrathecal Autologous Stem Cells — Patients will be stimulated with Granulocyte Colony Stimulating Factor (G-CSF) 5 times, harvest bone marrow and infused 8 to 10 mL of stem cells (CD34+) by intrathecal via.
  Other Names: Autologous Stem Cells Transplantation

SUMMARY:
The purpose of this study is to determine whether the plasticity of autologous intrathecal hematopoietic cells would improve the neurologic evolution of the pediatric patients with hypoxic/ischemic brain injury.

DETAILED DESCRIPTION:
There is accumulating evidence that shows that the placement of hematopoietic cells in the brain may increase growth-enhancing factors of axons and generate active neurons in the receptor. It has been found that after introducing hematopoietic cells in the subarachnoid space of the spinal cord, these cells may be transported through the cerebrospinal fluid and can be deliver more efficiently to the injured area, when compared to the intravenous route. Patients will be stimulated 4 times and then harvest the bone marrow. Bone marrow will be processed in order to obtain hematopoietic cells (CD34+) and minimize the erythrocytes amount. A inoculum of 5 to 10mL of stem cells will be infused intrathecally. Patients will be evaluated with the "Battelle Developmental Inventory" before the procedure and one and six months after that. An MRI will be performed before the procedure and six months after that.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypoxic/ischemic brain injury, with an between 1 month and 18 years, regardless the age at the time of injury, time post-injury, or previously received therapies, different from ours.

Exclusion Criteria:

* Patients with neurodegenerative or autoimmune diseases.
* Patients with active infection in any organ or tissue at the time of entering the study, the onset of stimulation with G-CSF or at the procedure.
* Patients who do not sign the informed consent form.

Elimination Criteria

* Patients with severe meningeal abnormalities at the time of procedure.
* Patients who did not attend subsequent assessments 30 and 180 days after the procedure.
* Patients who die from causes related to neurological disease within 180 days after procedure.
* Patients who are diagnosed with neurodegenerative or autoimmune diseases after the procedure.
* Patients who do not bear the proper stimulation process with Granulocyte Colony Stimulating Factor (G-CSF), either by misapplication, lack thereof, or severe adverse drug reaction.
* Patients choosing to leave the study.

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2009-07; Primary Completion 2010-04 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Score of "Battelle Developmental Inventory" | 30 days

SECONDARY OUTCOMES:
Score of "Battelle Developmental Inventory" | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Mancias-Guerra, MD, Principal Investigator — Hospital Universitario Dr. Jose E. Gonzalez; Arturo Garza-Alatorre, MD, Study Director — Hospital Universitario Dr. Jose E. Gonzalez; Laura N Rodriguez-Romo, MD, Study Chair — Hospital Universitario Dr. Jose E. Gonzalez
Locations (1):
- Hospital Universitario Dr. Jose E. Gonzalez, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Felling RJ, Snyder MJ, Romanko MJ, Rothstein RP, Ziegler AN, Yang Z, Givogri MI, Bongarzone ER, Levison SW. Neural stem/progenitor cells participate in the regenerative response to perinatal hypoxia/ischemia. J Neurosci. 2006 Apr 19;26(16):4359-69. doi: 10.1523/JNEUROSCI.1898-05.2006. PMID 16624956
- [Background] Glascoe FP, Byrne KE. The usefulness of the Battelle Developmental Inventory Screening Test. Clin Pediatr (Phila). 1993 May;32(5):273-80. doi: 10.1177/000992289303200504. PMID 7686835
- [Background] Berls AT, McEwen IR. Battelle developmental inventory. Phys Ther. 1999 Aug;79(8):776-83. No abstract available. PMID 10440664
- [Background] Levison SW, Rothstein RP, Romanko MJ, Snyder MJ, Meyers RL, Vannucci SJ. Hypoxia/ischemia depletes the rat perinatal subventricular zone of oligodendrocyte progenitors and neural stem cells. Dev Neurosci. 2001;23(3):234-47. doi: 10.1159/000046149. PMID 11598326
- [Background] Hayashi T, Iwai M, Ikeda T, Jin G, Deguchi K, Nagotani S, Zhang H, Sehara Y, Nagano I, Shoji M, Ikenoue T, Abe K. Neural precursor cells division and migration in neonatal rat brain after ischemic/hypoxic injury. Brain Res. 2005 Mar 15;1038(1):41-9. doi: 10.1016/j.brainres.2004.12.048. PMID 15748871
- [Background] Mehta T, Feroz A, Thakkar U, Vanikar A, Shah V, Trivedi H. Subarachnoid placement of stem cells in neurological disorders. Transplant Proc. 2008 May;40(4):1145-7. doi: 10.1016/j.transproceed.2008.03.026. PMID 18555135
- [Background] Goldman SA, Schanz S, Windrem MS. Stem cell-based strategies for treating pediatric disorders of myelin. Hum Mol Genet. 2008 Apr 15;17(R1):R76-83. doi: 10.1093/hmg/ddn052. PMID 18632701
- [Background] Eglitis MA, Mezey E. Hematopoietic cells differentiate into both microglia and macroglia in the brains of adult mice. Proc Natl Acad Sci U S A. 1997 Apr 15;94(8):4080-5. doi: 10.1073/pnas.94.8.4080. PMID 9108108
- [Background] Mezey E, Key S, Vogelsang G, Szalayova I, Lange GD, Crain B. Transplanted bone marrow generates new neurons in human brains. Proc Natl Acad Sci U S A. 2003 Feb 4;100(3):1364-9. doi: 10.1073/pnas.0336479100. Epub 2003 Jan 21. PMID 12538864
- [Background] Li Y, Chen J, Chen XG, Wang L, Gautam SC, Xu YX, Katakowski M, Zhang LJ, Lu M, Janakiraman N, Chopp M. Human marrow stromal cell therapy for stroke in rat: neurotrophins and functional recovery. Neurology. 2002 Aug 27;59(4):514-23. doi: 10.1212/wnl.59.4.514. PMID 12196642
- [Background] Gordon PH, Yu Q, Qualls C, Winfield H, Dillon S, Greene PE, Fahn S, Breeze RE, Freed CR, Pullman SL. Reaction time and movement time after embryonic cell implantation in Parkinson disease. Arch Neurol. 2004 Jun;61(6):858-61. doi: 10.1001/archneur.61.6.858. PMID 15210522
- [Derived] Mancias-Guerra C, Marroquin-Escamilla AR, Gonzalez-Llano O, Villarreal-Martinez L, Jaime-Perez JC, Garcia-Rodriguez F, Valdes-Burnes SL, Rodriguez-Romo LN, Barrera-Morales DC, Sanchez-Hernandez JJ, Cantu-Rodriguez OG, Gutierrez-Aguirre CH, Gomez-De Leon A, Elizondo-Riojas G, Salazar-Riojas R, Gomez-Almaguer D. Safety and tolerability of intrathecal delivery of autologous bone marrow nucleated cells in children with cerebral palsy: an open-label phase I trial. Cytotherapy. 2014 Jun;16(6):810-20. doi: 10.1016/j.jcyt.2014.01.008. Epub 2014 Mar 15. PMID 24642016
- [Derived] Mackie AR, Losordo DW. CD34-positive stem cells: in the treatment of heart and vascular disease in human beings. Tex Heart Inst J. 2011;38(5):474-85. PMID 22163120